CLINICAL TRIAL: NCT02836691
Title: Autonomic Nervous System Role in Uncontrolled ASTHMA and the Paucigranulocitic Phenotype
Acronym: ANASTHMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IIBSP-SNA-2015-87
Record Dates: First submitted 2016-05-05; First posted 2016-07-19 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Autonomic nervous system; Uncontrolled severe asthma; Paucigranulocitic asthma phenotype; Stress
MeSH Terms: conditions — Asthma | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EKG to Control subjects (Active Comparator): healthy controls without asthma or other respiratory disease.
  Interventions: Device: EKG (electrocardiogram)
- EKG monitoring Mild asthma (Active Comparator): The clinical grade of asthma is assessed in terms of the type of current asthma control (as GEMA Guide 4.0)
  Interventions: Device: EKG (electrocardiogram)
- EKG monitoring severe control asthma (Active Comparator): The clinical grade of asthma is assessed in terms of the type of current asthma control (as GEMA Guide 4.0)
  Interventions: Device: EKG (electrocardiogram)
- EKG monitoring severe uncontrolled asthma (Active Comparator): The clinical grade of asthma is assessed in terms of the type of current asthma control (as GEMA Guide 4.0)
  Interventions: Device: EKG (electrocardiogram)

INTERVENTIONS:
Device: EKG (electrocardiogram) — Analysis of the heart rate variability with an electrocardiogram with a commercial device adapted to asthmatic patients using 12 leads, a respiratory band and a pulseoximeter.

SUMMARY:
The autonomic nervous system (ANS) plays an important role in asthma, primarily through the parasympathetic (by the cholinergic pathway) promoting bronchoconstriction. Asthma is a chronic inflammatory disease, however, bronchoconstriction is not always caused by bronchial inflammation, as occurs in paucigranulocitic phenotype or noninflammatory asthma. The hypothesis of this project is based on the activation of the parasympathetic nervous system (PNS) would be involved in the pathogenesis of noninflammatory asthma (paucigranulocitic phenotype) and emotional stress and poor control of patients with severe asthma. To determine the ANS involvement in the pathogenesis of paucigranulocItic phenotype in asthma and correlate emotional stress, mediated by the ANS, with uncontrolled severe asthma. 30 asthmatics with different clinical severity (mild, severe controlled and uncontrolled severe) will be recruited , along with a control group of 10 healthy people. Descriptive variables, spirometry, inflammatory parameters (FeNO and inflammatory cell count in induced sputum), blood, saliva, urine and hair to obtain stress markers (glucose, copeptin, prolactin, cortisol) will be collected, and be supplied validated questionnaires of asthma control, quality of life and stress. For monitoring the response of the ANS will be done through an electrocardiogram, recording the heart rate variability (HRV). This analysis is carried out with the collaboration of engineers specialized in the characterization of cardiovascular signals for measuring the ANS.

DETAILED DESCRIPTION:
1. Role of the ANS in asthma

   For decades it's considered that the autonomic nervous system (ANS) plays an important role in the pathophysiology and symptomatology of asthma.

   The ANS had important functions besides regulating airway, such as bronchial smooth muscle tone, secretions, blood flow, microvascular permeability, also acts on migration and release of inflammatory mediators. This complex interaction between inflammation and neuronal control of airway, with effects on inflammatory mediators in neurotransmitters, modulates the inflammatory response (hypersecretion, edema and release of pro-inflammatory mediators as mast cell), through the activation of cholinergic reflex. Cholinergic neuronal pathway has a dominant effect on bronchoconstriction, and therefore represents an excellent therapeutic target. Anticholinergics reduce bronchial hyperresponsiveness to a wide range of bronchoconstriction agents, such as prostanoids, histamine, bradykinin, capsaicin, exercise or allergens.
2. ANS and non-inflammatory asthma (paucigranulocitic)

   In asthma can distinguish different inflammatory phenotypes, commonly typified by the presence of eosinophil's or neutrophils, and that can be performed through non invasive techniques of inflammometric such as exhaled nitric oxide and induced sputum. But it's not always bronchoconstriction mediated by bronchial inflammation. There is a significant proportion of patients with asthma, about 40% in those not objective bronchial inflammation, to that asthma is called noninflammatory asthma or paucigranulocitic phenotype, to proceed with normal levels of eosinophil's and neutrophils in sputum. The pathogenesis of the phenotype is not well defined, although suspected to be caused by strictly mechanical mechanisms diameter of the airway induced nervous stimulation. Among these mechanisms, the PNS could play an important role, however there are no studies that have evaluated the activation of the PNS in different clinical inflammatory disease phenotypes.
3. Control of asthma and stress Emotional stress affects the appearance and development of asthma by acting directly on the pathogenic mechanisms of airways, since states of great psychological stress have been associated with impaired adrenal sympathetic system and adrenal-pituitary-hypothalamic axis (APH). The argument that psychological stress influences the autonomic control of the airways is based primarily on the fact that many of the same autonomous mechanisms seem to play a role in asthma are involved in the activation and regulation of the physiological response to stress as chronic stress can alter the APH axis, cortisol secretion which is attenuated, leading to an increase in secretion of inflammatory cytokines.
4. Non-Invasive methods to measure the role of ANS Some author's suggest that the altered autonomic control of the caliber of airway in asthma can be reflected through a parallel change in heart rate (HR), as it is shown that in the asthmatic population are more likely to elevated resting heart rate compared to asthmatic population. Asthma and allergy has been associated with an increased activity of the PNS and asthma causes an elevation of heart rate variability (HRV), based on the measurement of basal parasympathetic tone. In fact, the authors asthma severity associated with greater impairment of HRV.

Therefore, evaluation of ANS is of great interest for diagnosis, prognosis and monitoring of this respiratory disorder. Direct evaluation of the PNS is infeasible or impractical in these situations. However, non-invasive evaluation of the PNS is proposed through the HRV according to the standards of measurement, physiological interpretation and clinical use of guides working group of the European Society and American Cardiology and Electrophysiology that are made through the electrocardiogram (ECG).

Ultimately, this research project aims to evaluate in a comprehensive manner the role it can play the ANS in the pathogenesis of asthma, namely the uncontrolled and non-inflammatory asthma severe asthma. The results of this study could provide new clues to understand why other mechanisms of asthma that do not pass through inflammatory. And therefore identification or further characterization of the role of ANS in the disease could generate preliminary evidence on which lay further research aimed at developing new molecules with anticholinergic capacity to treat asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged over 16 diagnosed with asthma (according to criteria GEMA 4.0). The diagnosis of asthma is assumed when the patient records stating suggestive previous symptoms of asthma with variable airflow obstruction (determined by spirometry or meter peak flow) or positive bronchodilator test (increase of 12% and 200 ml. of FEV1 after inhalation of a bronchodilator) or positive test to unspecific bronchoconstriction.

Exclusion Criteria:

* Asthma exacerbations a month before the visit
* Concomitance of other chronic respiratory diseases (bronchiectasis, fibrosis, etc.)
* Other important comorbidities in the opinion of investigators example: cardiovascular, endocrinological (especially diabetes, mental retardation, psychiatric or neurological disease relevant systemic inflammatory or immune disease

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | 2 years
  Comparison of heart rate variability (HRV) through an EKG among the group of non-inflammatory asthma (paucigranulocitic) with the rest of inflammatory phenotypes of severe asthma analyzed.

SECONDARY OUTCOMES:
Stress | 2 years
  Stress will be evaluated with validated questionnaires. Hospital Anxiety and Depression Scale (HADS)
Glucose (mg/dL) | 2 years
  Blood determination of glucose (mg/dl) as biomarker of emotional stress in patients with severe uncontrolled asthma.
copeptin (pmol/L) | 2 years
  Blood determination of copeptin (pmol/L) as biomarker of emotional stress in patients with severe uncontrolled asthma.
Prolactin (ng/mL) | 2 years
  Blood determination of prolactin (ng/mL) as biomarker of emotional stress in patients with severe uncontrolled asthma.
Salivary cortisol (ng/ml) | 2 years
  Salivary determination of cortisol (ng/ml) as biomarker of emotional stress in patients with severe uncontrolled asthma.
Salivary alpha-amylase U/L | 2 years
  Salivary determination of alpha-amylase U/L as biomarker of emotional stress in patients with severe uncontrolled asthma.
Urine cortisol (mcg/24h) | 24 hours
  Urine cortisol (mcg/24h) as biomarker of emotional stress in patients with severe uncontrolled asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Soto-Retes, physician, Principal Investigator — Santa Creu i Sant Pau Hospital
Locations (1):
- Lorena Soto-Retes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kaliner M, Shelhamer JH, Davis PB, Smith LJ, Venter JC. Autonomic nervous system abnormalities and allergy. Ann Intern Med. 1982 Mar;96(3):349-57. doi: 10.7326/0003-4819-96-3-349. PMID 6277221
- [Result] Barnes PJ. Neuroeffector mechanisms: the interface between inflammation and neuronal responses. J Allergy Clin Immunol. 1996 Nov;98(5 Pt 2):S73-81; discussion S81-3. PMID 8939180
- [Result] Gosens R, Bos IS, Zaagsma J, Meurs H. Protective effects of tiotropium bromide in the progression of airway smooth muscle remodeling. Am J Respir Crit Care Med. 2005 May 15;171(10):1096-102. doi: 10.1164/rccm.200409-1249OC. Epub 2005 Feb 1. PMID 15695490
- [Result] Peters SP, Kunselman SJ, Icitovic N, Moore WC, Pascual R, Ameredes BT, Boushey HA, Calhoun WJ, Castro M, Cherniack RM, Craig T, Denlinger L, Engle LL, DiMango EA, Fahy JV, Israel E, Jarjour N, Kazani SD, Kraft M, Lazarus SC, Lemanske RF Jr, Lugogo N, Martin RJ, Meyers DA, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Walter MJ, Wechsler ME, Chinchilli VM, Bleecker ER; National Heart, Lung, and Blood Institute Asthma Clinical Research Network. Tiotropium bromide step-up therapy for adults with uncontrolled asthma. N Engl J Med. 2010 Oct 28;363(18):1715-26. doi: 10.1056/NEJMoa1008770. Epub 2010 Sep 19. PMID 20979471
- [Result] Malerba M, Ragnoli B, Radaeli A, Tantucci C. Usefulness of exhaled nitric oxide and sputum eosinophils in the long-term control of eosinophilic asthma. Chest. 2008 Oct;134(4):733-739. doi: 10.1378/chest.08-0763. PMID 18842911
- [Result] Schleich FN, Manise M, Sele J, Henket M, Seidel L, Louis R. Distribution of sputum cellular phenotype in a large asthma cohort: predicting factors for eosinophilic vs neutrophilic inflammation. BMC Pulm Med. 2013 Feb 26;13:11. doi: 10.1186/1471-2466-13-11. PMID 23442497
- [Result] Douwes J, Gibson P, Pekkanen J, Pearce N. Non-eosinophilic asthma: importance and possible mechanisms. Thorax. 2002 Jul;57(7):643-8. doi: 10.1136/thorax.57.7.643. PMID 12096210
- [Result] Wright RJ. Exploring biopsychosocial influences on asthma expression in both the family and community context. Am J Respir Crit Care Med. 2008 Jan 15;177(2):129-30. doi: 10.1164/rccm.200710-1526ED. No abstract available. PMID 18165380
- [Result] Haldar P, Pavord ID. Noneosinophilic asthma: a distinct clinical and pathologic phenotype. J Allergy Clin Immunol. 2007 May;119(5):1043-52; quiz 1053-4. doi: 10.1016/j.jaci.2007.02.042. PMID 17472810
- [Result] Lehrer PM, Isenberg S, Hochron SM. Asthma and emotion: a review. J Asthma. 1993;30(1):5-21. doi: 10.3109/02770909309066375. PMID 8428858
- [Result] Wright RJ, Rodriguez M, Cohen S. Review of psychosocial stress and asthma: an integrated biopsychosocial approach. Thorax. 1998 Dec;53(12):1066-74. doi: 10.1136/thx.53.12.1066. PMID 10195081
- [Result] Kallenbach JM, Webster T, Dowdeswell R, Reinach SG, Millar RN, Zwi S. Reflex heart rate control in asthma. Evidence of parasympathetic overactivity. Chest. 1985 May;87(5):644-8. doi: 10.1378/chest.87.5.644. PMID 3987376
- [Result] Shah PK, Lakhotia M, Mehta S, Jain SK, Gupta GL. Clinical dysautonomia in patients with bronchial asthma. Study with seven autonomic function tests. Chest. 1990 Dec;98(6):1408-13. doi: 10.1378/chest.98.6.1408. PMID 2245682
- [Result] Garrard CS, Seidler A, McKibben A, McAlpine LE, Gordon D. Spectral analysis of heart rate variability in bronchial asthma. Clin Auton Res. 1992 Apr;2(2):105-11. doi: 10.1007/BF01819665. PMID 1638105
- [Result] Tokuyama K, Morikawa A, Mitsuhashi M, Mochizuki H, Tajima K, Kuroume T. Beat-to-beat variation of the heart rate in children with allergic asthma. J Asthma. 1985;22(6):285-8. doi: 10.3109/02770908509087111. PMID 4077809
- [Result] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210